CLINICAL TRIAL: NCT05159531
Title: Virtual PrEP: Rendering PrEP Delivery More Efficient Using an mHealth Intervention and TAF/FTC
Brief Title: Virtual PrEP: Rendering PrEP Delivery More Efficient
Acronym: VPrEP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: Unity Health Toronto (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CTN 332
Record Dates: First submitted 2021-11-03; First posted 2021-12-16 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: HIV Infections
Keywords: HIV; PrEP; HIV prevention
MeSH Terms: conditions — HIV Infections | interventions — emtricitabine tenofovir alafenamide; Standard of Care

STUDY DESIGN:
Intervention Model Description: 1:1 open-label RCT using a AB:BA crossover design, comparing the standard of care to an mHealth-based model of care for TAF/FTC PrEP delivery over 72 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard model of care (Experimental): Delivery of PrEP care through the local standard of care.
  Interventions: Drug: PrEP; Other: Standard of Care
- mHealth model of care (Active Comparator): Delivery of PrEP care through the Freddie® mobile Health (mHealth) platform.
  Interventions: Drug: PrEP; Other: mHealth Model of Care

INTERVENTIONS:
Drug: PrEP — Participants will receive Descovy® 200/25mg 1 tablet once daily for 72 weeks.
  Other Names: Descovy® 200/25mg (DIN= 02454424); TAF/FTC; tenofovir alafenamide/emtricitabine
Other: mHealth Model of Care — Freddie® allows for asynchronous contact between patients and care providers, meaning that it does not require both groups to be connected in real time, instead allowing communication over a number of days.
  Other Names: GoFreddie®
  Arms: mHealth model of care
Other: Standard of Care — Delivery of PrEP care through the local standard of care
  Other Names: PrEP standard of care
  Arms: Standard model of care

SUMMARY:
Gay, bisexual and other men who have sex with men (GBM) account for over half of new HIV infections in Canada each year, and have a 131-fold higher risk of HIV than other Canadian men. HIV pre-exposure prophylaxis (PrEP) using regular oral tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) or tenofovir alafenamide/emtricitabine (TAF/FTC) is an effective and safe HIV prevention option.

Despite growing interest, awareness and willingness to use PrEP there has been numerous challenges to the broader rollout of PrEP. This study will address some of these challenges by assessing participant satisfaction,feasibility and clinical outcomes associated with a web-based mobile health (mHealth) model of care for daily oral TAF/FTC PrEP compared to standard of care delivery of TAF/FTC PrEP in Canadian GBM/TGW, in the era of COVID-19.

The ultimate goal of this study is to provide a scalable model for remote PrEP delivery that minimizes the need for in-person interactions; respects guideline recommendations regarding how to optimally monitor patients; and is attractive to both patients and providers.

This study is a 1:1 open-label, pragmatic randomized controlled trial using a AB:BA crossover design, comparing the standard of care to an mHealth based model of care (Freddie® ) for TAF/FTC PrEP delivery over 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported gay, bisexual or other man who has sex with men (inclusive of transgender men) or transgender woman
2. Age ≥16
3. HIV seronegative, as documented by a 4th generation HIV antigen/antibody combination test performed within 14 days of baseline
4. No symptoms of acute HIV seroconversion (fever, myalgias, arthralgias, malaise, headache, rash, pharyngitis and/or diarrhea that is otherwise unexplained)
5. Meets clinical criteria for PrEP according to the prescribing clinician. Patients can be enrolled into the study regardless of whether they will be newly initiating PrEP, or are already receiving PrEP; those already receiving PrEP can be using any regimen (eg. daily TDF/FTC, on-demand TDF/FTC, daily TAF/FTC) as long as they are willing to transition to the study regimen of daily, oral TAF/FTC.
6. eGFR >30ml/min
7. Has adequate access to the internet to permit use of the mHealth platform
8. Adequate facility in English to communicate with their provider

Exclusion Criteria:

1. Known hypersensitivity/allergy to TAF/FTC
2. Actively participating in another interventional trial related to the delivery of PrEP or sexual health-related care
3. Being unwilling or unable to perform self-collected pharyngeal and/or rectal swabs as part of routine PrEP care
4. Potential to become pregnant
5. Currently living in, or planning to move to a location that would render standard of care or ad hoc in-person visits to the study site impractical during the study period.

Min Age: 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Self-reported gay, bisexual or other man who has sex with men or transgender woman
Enrollment: 2 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
'Final Visit Questionnaire' will be used to determine participants' stated preference for either the standard of care or the mHealth-based model of care. | 72 weeks
  The primary outcome will be defined using the response to the following question:
  "During this study, your PrEP care was provided through the Freddie platform for part of the study period, and through your clinic's standard procedures for part of the study period. Which of these did you prefer?"

SECONDARY OUTCOMES:
Study visit attendance will be used to compare the number of missed visits by model of care | 72 weeks
  Measured by study visit attendance (defined as: occasions on which the patient and provider fail to connect for a quarterly follow-up in the pre-planned fashion)
Quantity of missing laboratory questionnaires will be used to compare the number of missed laboratory evaluations by model of care. | 72 weeks
  Missed laboratory evaluations (secondary outcome B) will be defined as any occasion on which a participant fails to complete their clinically indicated laboratory tests (HIV serology, STI screening, creatinine) by the end of the 9th week of each 12-weekly follow-up cycle.
Interview administered questionnaires will be used to comparison of the average amount of participant time required for PrEP follow-up activities by model of care | 72 weeks
  Measure of time required for PrEP follow-up activities per quarter will be calculated as the sum (in minutes) of all time spent by the participant on activities related to receiving PrEP care per 12-week follow-up interval, as reported by the participant during study interviews.
Questionnaires administered to clinicians will be used to compare of the average amount of clinician time required for PrEP follow-up by activities per model of care | 72 weeks
  Measured by total number of minutes spent by the clinician on activities related to delivering PrEP care per 12-week follow-up interval.
Study visit attendance will be followed to compare of the total number of participant visits by model of care | 72 weeks
  measured from study visit attendance
PrEP adherence questionnaire administered at week 36 and 72 will be used to determine PrEP adherence. | 72 weeks
  PrEP adherence refers to the degree to which participants take their daily TAF/FTC as prescribed. PrEP adherence questionnaire will include questions of the number of days per week on which PrEP was taken.
Dried blood spot will be collected at week 36 and 72 will be used to determine PrEP adherence. | 72 weeks
  PrEP adherence refers to the degree to which participants take their daily TAF/FTC as prescribed. Samples will be analyzed for drug levels as this outcome is mapped onto pharmacokinetic outcomes.
Hair Samples will be collected at week 36 and 72 will be used to determine PrEP adherence. | 72 weeks
  PrEP adherence refers to the degree to which participants take their daily TAF/FTC as prescribed. Samples will be analyzed for drug levels as this outcome is mapped onto pharmacokinetic outcomes.
Participant visit logs will be used to assess retention in PrEP care by model of care. | 72 weeks
  Measurement of patients' continued engagement in PrEP care, regardless of whether continuing to take PrEP medication.
Interview administered questionnaires will be used to qualitatively learn about the preferences of patients and providers about the mHealth model of care. | 72 weeks
  Questions assessing pros and cons of each model of care will allow for participants to provide insight about preferences in PrEP care models.
Satisfaction questionnaires will be used to compare participant satisfaction with their PrEP care by model of care. | 72 weeks
  Measured by questionnaire responses at weeks 4, 12, 36, 48, 60 and at final study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Darrell HS Tan, MD,FRCPC,PhD, Principal Investigator — Unity Health Toronto; Kevin Woodward, MD,FRCPC, Principal Investigator — Hamilton PrEP Clinic
Locations (5):
- Canada (5):
  - Sexually Transmitted Infection (STI) Clinic, Calgary, Alberta
  - Nine Circles, Winnipeg, Manitoba
  - Hamilton PrEP Clinic, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Maple Leaf Research, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No